CLINICAL TRIAL: NCT07020650
Title: The Effectiveness of Carbonate Apatite Bone Graft for Alveolar Ridge Preservation: A Clinical, Radiographic, and Histomorphometric Study
Brief Title: The Effectiveness of Carbonate Apatite Bone Graft for Alveolar Ridge Preservation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, Department of Periodontics and Oral Medicine, School of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00267966
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healing Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Synthetic bone (Experimental): Bone graft with carbonate apatite (Cytrans Granules)
  Interventions: Procedure: Socket preservation
- Allograft (Active Comparator): Bone graft with allograft (Puros)
  Interventions: Procedure: Socket preservation
- Xenograft (Experimental): Bone graft with xenogeneic plug (BioOss)
  Interventions: Procedure: Socket preservation

INTERVENTIONS:
Procedure: Socket preservation — After tooth extraction, the socket will be filled with a collagen plug and bone graft.

SUMMARY:
This study will examine whether the use of synthetic carbon apatite bone graft material will lead to more bone formation compared to human derived allograft and bovine derived xenograft material.

DETAILED DESCRIPTION:
Bone grafts are commonly placed to increase the amount of bone right after tooth extraction and prepare the site for future dental implant placement.

45 patients requiring a tooth extraction will be recruited and randomized to receive either allograft, xenograft, or synthetic bone grafting.

ELIGIBILITY:
Inclusion criteria:

* Age between 20 and 80 years old
* Patients requiring tooth extraction (incisors, canines, and premolars) due to caries, periodontal disease, tooth fracture, or unrestorable condition.
* Extraction sockets must be infection-free with dehiscence less than 5mm.
* Patients interested in implant placement after tooth extraction.

Exclusion criteria:

* Known allergies or hypersensitivities to medications related to the study (e.g., chlorhexidine)
* Hematologic disorders or blood dyscrasias.
* Active infectious diseases.
* Liver or kidney dysfunction/failure.
* Uncontrolled diabetes (i.e., HbA1c > 8).
* Undergoing active cancer treatment, including chemotherapy or radiotherapy within the last 12 months from the procedure.
* Use of medications affecting bone healing (e.g., bisphosphonates, long-term anti-inflammatory medications).
* Metabolic bone diseases affecting bone healing, such as osteoporosis (self-reported).
* Pregnant or lactating women (self-reported).
* Current smokers of 10 or more cigarettes per day and former smokers who quit less than 10 years ago (self-reported).
* Poor oral hygiene.
* Presence of fenestration defects equal to or greater than 5mm.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical alveolar ridge dimension changes | 4 months
  Clinically measured alveolar ridge dimension changes in mm

SECONDARY OUTCOMES:
Histological bone density | 4 months
  Histomorphometry
Presence of bone turnover proteins | 4 months
  Immunohistochemistry
Alveolar volumetric changes following tooth extraction | 4 months
  Digitally measured alveolar ridge changes in mm^3 using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS,MSD,PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No